CLINICAL TRIAL: NCT01420887
Title: Preservation of Joint Function Using Postoperative Continuous Passive Motion (CPM) A Pilot Study
Acronym: CPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shawn W. O'Driscoll, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-000601
Record Dates: First submitted 2011-07-13; First posted 2011-08-22 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Elbow Injury
Keywords: CPM; elbow joint surgery; continuous passive motion; Recovery after surgery to restore elbow motion
MeSH Terms: conditions — Elbow Injuries | interventions — Motion Therapy, Continuous Passive; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Passive Motion (Experimental): Subjects randomized to CPM therapy.
  Interventions: Procedure: Continuous Passive Motion
- Physical Therapy (Active Comparator): Subjects randomized to physical therapy.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Continuous Passive Motion — Continuous passive motion.
  Arms: Continuous Passive Motion
Procedure: Physical Therapy — Physical therapy.
  Arms: Physical Therapy

SUMMARY:
This pilot study is designed to determine if the rehabilitative benefits of continuous passive motion (CPM) will help preserve/restore the joint function and significantly improve the rate of recovery of patients after the surgical release of elbow contractures better than standard physiotherapy and static splinting.

DETAILED DESCRIPTION:
Elbow stiffness and reduced motion commonly occur after elbow injury or surgery. With traumatic injuries to the elbow, contractures are a common complication. Indeed, they are expected in most cases. For patients with these injuries who are otherwise healthy, active and require the restoration of full function in order to return to their previous level of activity/work, this reduced motion can be especially problematic and even debilitating. The investigators have found and published that most patients treated with postoperative Continuous Passive Motion following surgical repair of their stiffness have been able to recover all or nearly all of their prior elbow mobility and function. Though CPM has been in clinical use for decades, a prospective randomized clinical trial has never been published proving its effectiveness. The investigators believe and intend to show in this study that the rehabilitative benefits of continuous passive motion (CPM) will help preserve/restore the joint function and significantly improve the rate of recovery of patients after stiffness is surgically repaired. Specific Aim 1: To demonstrate that postoperative use of CPM enhances tissue healing and hastens recovery following surgical release of elbow contracture. Specific Aim 2: To demonstrate that postoperative use of CPM improves ultimate function following surgical release of elbow contracture. Specific Aim 3: To demonstrate that CPM is a cost-efficient treatment following surgical release of elbow contracture. Study Design: 50 patients who require arthroscopic contracture release, will be randomly assigned to one of two postoperative treatment groups: Experimental - CPM and Control - Physical Therapy. Participants of this study will be followed for 12 months postoperatively. Throughout this 12 month period the impact/effectiveness of CPM vs Physical Therapy will be evaluated by assessing functional status, pain, mobility, general health related quality of life, utility, and societal cost-effectiveness. In line with the mission of the National Institute of Arthritis and Musculoskeletal and Skin Diseases, this study will help anyone with elbow injuries that result in stiffness and loss of motion. Such a study has the advantage of being highly translational with the potential to have an immediate impact on patient treatment and care. The findings from this study will be able to help patients immediately and ensure that the principals of Evidence Based Medicine are applied to patients with these types of elbow injuries and that they receive the treatment they need for the best possible recovery based on hard evidence and scientific facts.

ELIGIBILITY:
Inclusion Criteria:

To be included, each patient must meet ALL of the following:

1. Lack of elbow flexion and/or extension, with or without pain.
2. The contracture must have been present for at least six months and failed to respond to non-surgical treatment.
3. Surgery to be performed will be arthroscopic capsulectomy or osteocapsular arthroplasty with removal of heterotopic ossification as necessary

Exclusion Criteria:

1. Contraindication to use of CPM or regional brachial plexus block, such as bleeding diathesis, use of anticoagulants or severe restriction in shoulder range of movement.
2. Progressive or recalcitrant neuropathy or neuritis, except for isolated intermittent ulnar neuritis.
3. Pre-existing factors that might limit ability to completely participate in rehabilitations such as neuromuscular or psychosocial condition.
4. Progressive or recurrent contracture due to inflammatory disease such as rheumatoid arthritis, juvenile idiopathic arthritis or chondrolysis.
5. Altered anatomy that might limit elbow motion, independent of the condition being treated, such as dysplasia, malunion, osteonecrosis, and congenital deformity.
6. A reasonable restoration of motion and function cannot be expected.
7. Inadequate postoperative regional anesthesia
8. Intra-operative or postoperative complication that could affect outcome
9. Injury or disease in the postoperative period that could affect elbow function
10. Not possible to have postoperative physical therapy appointment
11. Significant portion of the procedure performed in an open manner
12. Women that know they are pregnant or breastfeeding
13. Current or prior septic arthritis

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-18 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Recurrence of elbow contracture | 1 year
  There will be an 80% statistical power to detect a difference of 2 points in the pre-surgery to post-surgery change in VAS pain between subjects in the two study arms. Similarly, there will be an 80% power to detect a difference of 16 degrees in the pre-surgery to post-surgery change in total arc of motion between the two study groups. There will be 80% power to detect a difference of at least 9 points on the pre-surgery to post-surgery difference in the DASH score.

SECONDARY OUTCOMES:
Subsequent injury or disease of the affected elbow | 1 year
  There will be an 80% statistical power to detect a difference of 2 points in the pre-surgery to post-surgery change in VAS pain between subjects in the two study arms. Similarly, there will be an 80% power to detect a difference of 16 degrees in the pre-surgery to post-surgery change in total arc of motion between the two study groups. There will be 80% power to detect a difference of at least 9 points on the pre-surgery to post-surgery difference in the DASH score.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn O Driscoll, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials